CLINICAL TRIAL: NCT04423679
Title: The Selfie Study- Assessing Novel Markers for Cervical Cancer Screening From Self-collected Samples
Acronym: SELFIE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: George Washington University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nicole Chappell, Principle Investigator, George Washington University
Other Study IDs: NCR191015
Record Dates: First submitted 2020-05-18; First posted 2020-06-09 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Human Papilloma Virus; Cervical Cancer; CIN 2/3
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIN2+: Cases of cervical precancer will include women diagnosed with cervical intraepithelial grades 2 or 3 (CIN2/3) or adenocarcinoma in situ (AIS). If any women are diagnosed with cancer in the study, they will be included in this group.
  Interventions: Device: Evalyn Brush
- < CIN2: Non-cases will include those with <CIN2 on colposcopy/biopsy and women who did not have an indication for colposcopy (because of a negative screening test).
  Interventions: Device: Evalyn Brush

INTERVENTIONS:
Device: Evalyn Brush — a standard brush-based cervicovaginal self-collection device

SUMMARY:
Cervical cancer is primarily caused by Human Papillomaviruses (HPV). Testing for HPV in cervical samples is now an option for cervical cancer screening. HPV can also be tested from self-collected samples which may help to improve access to screening, since it does not require a doctor visit. However, many women will test positive for HPV who are not at high risk for cervical cancer. Therefore, additional ("triage") tests are needed to determine which women testing HPV-positive require additional clinical workup. For self sampling, a triage test that could be measured from the same initial sample without requiring a follow-up visit to the doctor would be an ideal strategy. The purpose of this study is to determine whether a new HPV test that measures changes in HPV DNA can be used to triage HPV-positive women using self collected samples. This study will enroll 1,000 women who are undergoing cervical cancer screening at the George Washington University. Women will be asked to take a self-collected sample prior to their clinic visit. The investigators will evaluate the clinical accuracy of the new HPV triage test in self-collected samples and compare the accuracy of the test in samples collected by the clinician.

DETAILED DESCRIPTION:
Worldwide, cervical cancer remains the fourth most common cancer and fourth leading cause of cancer deaths among women, with the greatest burden occurring in low-resource settings that lack effective screening and treatment. Even in the United States (U.S.), where Pap cytology screening has resulted in dramatic declines in cervical cancer incidence and mortality, thousands of new cases and related-deaths still occur every year, most commonly among underserved women who face barriers to accessing screening and/or treatment. The recent implementation of human papillomavirus (HPV) DNA testing as a primary strategy for cervical cancer screening has the potential to alleviate these disparities by improving the sensitivity for cervical precancer detection compared to Pap cytology, while providing greater long term reassurance following a negative HPV test. Moreover, HPV testing can be successfully performed on self-collected specimens, offering the possibility of expanding access to cervical cancer screening among hard-to-reach, underserved women.

Despite the many advantages of primary HPV screening, the current challenge is optimizing triage testing to determine who among the many women testing HPV positive are at high-risk and require immediate colposcopy referral or treatment, while avoiding unnecessary harms among women at low-risk. A molecular triage test that can be conducted from the same primary screening sample (i.e., reflex testing) is particularly attractive for both high-and low-resource settings, particularly if it works from self-collected samples. Previously, DNA methylation of candidate host cell genes has been evaluated in self-collected samples and achieved acceptable performance for triage of HPV-positive women. In studies using clinician collected samples, there is a suggestion that methylation of carcinogenic HPV genotypes has better clinical performance (higher sensitivity/specificity) compared to host gene methylation; however, HPV methylation has not been evaluated in self-collected specimens. Because HPV DNA is present in only a small subset of infected cells in the lower genital tract, particularly in cervical precancers, it is likely that the signal-to noise ratio in self-collected samples is better for HPV compared to host gene methylation, resulting in improved specificity for cervical precancer detection. Evaluating the feasibility of HPV DNA methylation testing from self-collected samples is essential for determining the extent to which this assay can address the critical need for HPV triage in high- and low resource settings. In collaboration with the Cancer Genome Research Laboratory, a high-throughput, low-cost next-generation bisulfite sequencing assay that detects methylation of the 12 most carcinogenic HPV genotypes has been developed. Further, this assay includes a panel of host genes, including those that have been previously evaluated in self-collected specimens. The proposal is to test this assay in paired self and clinician-collected samples from 1,000 women enrolled in an ongoing prospective study of women undergoing cervical cancer screening and colposcopy at the George Washington University (GWU). The hypothesis is that HPV and host DNA methylation will show non-inferior sensitivity and specificity for detection of cervical precancer in self-collected compared to clinician-collected samples and that HPV methylation will have higher absolute specificity compared to host methylation in both sample types.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 30-69
* Undergoing cervical cancer screening, diagnostic procedure (colposcopy), or treatment (LEEP)

Exclusion Criteria:

* Pregnancy
* History of Cervical Cancer
* Prior hysterectomy
* Inability to provide informed consent

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women undergoing routine screening with Pap cytology and HPV testing or colposcopy at the George Washington University (GWU). From this population, a representative subset of 1000 women for self-sampling and methylation testing (400 cases and 600 controls). Most controls will come from the screening population, where we expect 85% to have negative HPV and cytology results. The majority of cases will come from the colposcopy referral population. Cases of cervical precancer will include women diagnosed with cervical intraepithelial grades 2 or 3 (CIN2/3) or adenocarcinoma in situ (AIS). If any women are diagnosed with cancer in the study, they will be included in the case group (CIN2+); however, we will also perform sensitivity analyses excluding these women. Non-cases will include those with less than CIN2 on colposcopy/biopsy and women who did not have an indication for colposcopy (because of negative screening).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluating the relative sensitivity and specificity of HPV methylation testing from collected samples | Up to 24 months
  Evaluate the relative sensitivity and specificity of HPV methylation testing from self-collected compared to clinician-collected samples for detection of cervical precancer.
Evaluating the relative sensitivity and specificity of host gene methylation testing from collected samples | Up to 24 months
  Evaluate the relative sensitivity and specificity of host gene methylation testing from self-collected compared to clinician-collected samples for detection of cervical precancer.
Comparing the absolute sensitivity and specificity of HPV versus host gene methylation testing | Up to 24 months
  Compare the absolute sensitivity and specificity of HPV versus host gene methylation testing for the detection of cervical pre-cancer in both self-collected and clinician-collected samples

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No